CLINICAL TRIAL: NCT02517437
Title: Novel Combination of Suprascapular & Axillary Nerve Blocks Versus Conventional Interscalene Brachial Plexus Block for Pain Relief Following Shoulder Surgery: A Multi-centre Randomized, Patient & Assessor Blinded, Non-inferiority Trial
Brief Title: Suprascapular and Axillary Blocks Versus Interscalene Block for Shoulder Surgery
Acronym: PASS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REB14-8557-A
Record Dates: First submitted 2015-07-20; First posted 2015-08-07 (Estimated); Last update posted 2018-05-31 (Actual); Status verified 2018-03

CONDITIONS: Shoulder Pain
MeSH Terms: conditions — Shoulder Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Suprascapular & axillary blocks (Active Comparator): Suprascapular and axillary blocks.
  Interventions: Drug: Suprascapular & axillary blocks
- Interscalene block (Active Comparator): Interscalene block.
  Interventions: Drug: Interscalene block

INTERVENTIONS:
Drug: Suprascapular & axillary blocks — After infiltration with 1 mL of 1% lidocaine, local anesthetics (20 mL of 0.5% ropivacaine) will then be injected in 5 mL aliquots to achieve circumferential spread around the nerve.The axillary nerve block will be performed next in the posterior aspect of the operative arm. The neurovascular bundle encompassing the humeral artery, posterior circumflex artery, and axillary nerve is visualized in the lateral edge of the quadrangular space, deep to the deltoid muscle, inferior to the teres minor muscle, and superior to the triceps tendon. After infiltration with 1 mL of 1% lidocaine, local anesthetics (20 mL of 0.5% ropivacaine) will then be injected in 5 mL aliquots after negative aspiration to achieve circumferential spread around the bundle.
  Other Names: Suprascapular and axillary blocks
  Arms: Suprascapular & axillary blocks
Drug: Interscalene block — After sterile skin preparation with chlorhexidine and infiltration with 1 mL of 1% lidocaine, a 5 cm 22 G insulated needle is then inserted and local anesthetic solution (20 mL of 0.5% ropivacaine) will be injected in 5 mL aliquots after negative aspiration for blood to achieve spread posterior to or between the C5 and C6 nerve roots.
  Arms: Interscalene block

SUMMARY:
The purpose of this study is to determine whether the combination of suprascapular and axillary nerve blocks is non-inferior to the conventional interscalene block (ISB) in providing pain relief during the first postoperative day to adult healthy patients (age > 18) undergoing ambulatory shoulder surgery.

DETAILED DESCRIPTION:
Study Hypothesis:The pain relief provided by a combination of suprascapular and axillary nerve blocks is non-inferior to that produced by the conventional interscalene block during the first 24hours postoperatively in adult patients undergoing ambulatory shoulder surgery.

Intervention and Comparator: Consented patients will be randomized to receive either pre-operative ISB (plus sham SAB with subcutaneous saline), or SAB (plus sham ISB). Both groups will receive general anesthesia for surgery.

Primary Aim: To demonstrate non-inferiority of pain relief produced by the combination treatment compared to the conventional treatment by comparing the area under the curve of the postoperative pain scores plot over time during the first 24 hours postoperatively.

Secondary Aims: There are four secondary aims, covering efficacy (analgesia) and safety: rest pain, quality of recovery, safety, other pain relief indicators.

Design There will be a multi-centre, prospective, randomized, patient and assessor blinded, two-arm, parallel-group, 1:1 allocation ratio, placebo-controlled, non-inferiority clinical trial comparing the effect of SAB treatment to conventional ISB treatment on pain relief during the first postoperative 24 hours in patients undergoing ambulatory shoulder surgery under general anesthesia.

Methods Study participants

The target population will be adult patients (age > 18) presenting for outpatient (same day surgery) unilateral arthroscopic or open shoulder surgery. Eligible surgical procedures are:

* Shoulder arthroscopy
* Shoulder instability procedures

  1. Superior labrum anterior posterior repair (SLAP)
  2. Rotator cuff repair
  3. Bankart repair
* Acromioplasty

Study centres The trial will be conducted at the two academic medical centres in Toronto where ambulatory shoulder surgery is routinely performed: Toronto Western Hospital (TWH),and Women's College Hospital (WCH).

Preoperative management Unless allergic, all patients will receive acetaminophen 1 gr and celecoxib 400 mg orally with sips of water one hour prior to surgery. All blocks will be performed in the block room one hour before surgery.

Suprascapular and axillary nerve blocks (SAB group) Patients allocated to the suprascapular and axillary nerve block combination (SAB group) will receive these blocks in the sitting position. The shoulder will be in the neutral position but rotated 45 degrees inward and the elbow flexed at 90 degrees while the hand rests on the knees. The suprascapular nerve will be blocked as it branches from the superior trunk.78After sterile skin preparation with chlorhexidine, a linear array transducer (6-13 MHz, Sonosite M-Turbo) probe protected by a 3M Tegaderm® dressing or a sterile sheath is placed in the transverse plane to visualize C5 and C6 roots in the interscalene groove. These roots are then traced distally to where they coalesce to form the superior trunk. The suprascapular nerve is then identified and as it emerges from the superior trunk, under the deep cervical fascia and superficial to the middle scalene muscle. After infiltration with 1 mL of 1% lidocaine, a 5 cm 22 G insulated needle (B. Braun Medical Inc., Bethlehem, PA, USA) is inserted in line with the probe in a lateral-to-medial orientation towards the nerve. Local anesthetics (20 mL of 0.5% ropivacaine) will then be injected in 5 mL aliquots after negative aspiration for blood to achieve circumferential spread around the nerve.

The axillary nerve block will be performed next in the posterior aspect of the operative arm. The US transducer is placed in the longitudinal plane, parallel to the long axis of the humerus shaft and approximately 2cm below the postero-lateral part of the acromion on the posterior aspect of the arm. (Figure 1) The neurovascular bundle encompassing the humeral artery, posterior circumflex artery, and axillary nerve is visualized in the lateral edge of the quadrangular space, deep to the deltoid muscle, inferior to the teres minor muscle, and superior to the triceps tendon. After infiltration with 1 mL of 1% lidocaine, the 22G needle is inserted in line with the probe in a caudad orientation towards the bundle. Local anesthetics (20 mL of 0.5% ropivacaine) will then be injected in 5 mL aliquots after negative aspiration to achieve circumferential spread around the bundle.

Finally, to maintain patient blinding, sham ISB block will be performed in the semi-sitting position using a 25G needle to inject 1 mL of lidocaine 1% subcutaneously.

Interscalene block (ISB group) Local anesthetic solution (20 mL of 0.5% ropivacaine) will be injected in 5 mL aliquots after negative aspiration for blood to achieve spread posterior to or between the C5 and C6 nerve roots. Subsequently, patients will receive sham SAB performed in the sitting position using a 25G needle to inject 1 mL of lidocaine 1% subcutaneously.

Block assessment Assessment of sensory block onset to confirm block success is done by the research assistant doing the blocks every 5 minutes, for 30 minutes, with a blunt 22G needle applied to skin, by comparing to the contralateral upper extremity.

General anesthesia All patients will receive a standardized general anesthetic.

Postoperative management Discharged patients will receive a prescription for Tylenol #3® as needed, or Percocet® if intolerant to codeine.

Two-week follow-up A study follow-up phone call will be arranged to specifically assess any potential block-related neurologic symptoms such as pain, paresthesia, dysesthesia, sensory loss, motor power weakness. Patients found to have such symptoms will be offered a referral to the chronic pain clinic at TWH for assessment and management.

Data collection The study coordinators of the participating sites will use a paper-based case report form (CRF) prepared by the principal investigator for documentation of outcome results. Subject confidentiality will be maintained by using a study ID (not related to name, or date of birth) on all CRFs.

Sample Size Investigators aim to enroll a total of 65 patients per group, or a total of 130 patients. Based on the annual number of shoulder surgeries performed at each centre, the researchers plan to recruit 45 patients at TWH, and another 85 patients at WCH.

Source Data Verification: Patient Electronic Record

Quality Assurance & Data Checks: N/A

ELIGIBILITY:
Inclusion Criteria:

* Consented, English-speaking, adult patients (age > 18)
* American Society of Anesthesiologists (ASA) classification I-III
* BMI ≤ 30 kg/m2

Exclusion Criteria:

* Total shoulder arthroplasty or clavicular surgery (ISB does not provide sufficient pain relief)
* Known broncho-pulmonary or phrenic pathology compromising respiratory function
* Contra-indication to nerve blocks e.g., infection, bleeding diathesis, allergy to local anesthetics
* Existing chronic pain disorders or history of use of ≥ 30mg oxycodone or equivalent per day
* Pre-existing neurological deficits or peripheral neuropathy involving the operative upper extremity
* Contraindication to any component of multi-modal analgesia (acetaminophen, non-steroidal anti-inflammatory medications, oral opioid analgesics)
* Pregnancy or any significant psychiatric conditions that may affect patient assessment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2015-08; Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Postoperative pain severity | 1st post-operative 24 hours
  Numeric rating scale (NRS) scores will be evaluated by blinded study coordinators who are not involved in patient care.

SECONDARY OUTCOMES:
Rest pain at additional time points | 0, 6, 12, 18, and 24 hours postoperatively
Quality of Recovery (QoR) | 24 hours
  The impact of surgical and anesthetic interventions on perioperative quality of life and ability to resume routine life activities will be assessed using the Quality of Recovery (QoR) tool. The QoR-15 scale is a patient-based outcome measure in the form of a 15-item validated questionnaire.

OTHER OUTCOMES:
Hemodynamic side effect | 24 hours
  Hemodynamic side effects, defined as occurrence of bradycardia or hypo-tension.
Block success | 24 hours
  Block success is defined as complete sensory block over the deltoid.
Procedural complications | during or just after block.
  Procedural complications are defined as occurrence of intravascular injection, local anesthetic systemic toxicity, hematoma, pneumothorax, epidural spread, and Horner's syndrome

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Chan, MD, Principal Investigator — Toronto Western Hospital, University Health Network, University of Toronto; Faraj Abdallah, MD, Principal Investigator — St. Michael's Hospital, University of Toronto; Richard Brull, MD, Principal Investigator — Women's College Hospital, University of Toronto
Locations (2):
- Canada (2):
  - Women's College Hospital, Toronto, Ontario
  - Toronto Western Hopspital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Yes
publication

REFERENCES:
- [Background] Stark PA, Myles PS, Burke JA. Development and psychometric evaluation of a postoperative quality of recovery score: the QoR-15. Anesthesiology. 2013 Jun;118(6):1332-40. doi: 10.1097/ALN.0b013e318289b84b. PMID 23411725
- [Background] Voogd AC, Ververs JM, Vingerhoets AJ, Roumen RM, Coebergh JW, Crommelin MA. Lymphoedema and reduced shoulder function as indicators of quality of life after axillary lymph node dissection for invasive breast cancer. Br J Surg. 2003 Jan;90(1):76-81. doi: 10.1002/bjs.4010. PMID 12520579
- [Background] Peintinger F, Reitsamer R, Stranzl H, Ralph G. Comparison of quality of life and arm complaints after axillary lymph node dissection vs sentinel lymph node biopsy in breast cancer patients. Br J Cancer. 2003 Aug 18;89(4):648-52. doi: 10.1038/sj.bjc.6601150. PMID 12915872
- [Background] Lo IK, Litchfield RB, Griffin S, Faber K, Patterson SD, Kirkley A. Quality-of-life outcome following hemiarthroplasty or total shoulder arthroplasty in patients with osteoarthritis. A prospective, randomized trial. J Bone Joint Surg Am. 2005 Oct;87(10):2178-85. doi: 10.2106/JBJS.D.02198. PMID 16203880
- [Background] Gutierrez DD, Thompson L, Kemp B, Mulroy SJ; Physical Therapy Clinical Research Network; Rehabilitation Research and Training Center on Aging-Related Changes in Impairment for Persons Living with Physical Disabilities. The relationship of shoulder pain intensity to quality of life, physical activity, and community participation in persons with paraplegia. J Spinal Cord Med. 2007;30(3):251-5. doi: 10.1080/10790268.2007.11753933. PMID 17684891